CLINICAL TRIAL: NCT03279913
Title: NEUROFEEDSTIM : Therapeutic Use of Neurofeedback in Depression in Association With TMS
Acronym: NEUROFEEDSTIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 35RC16_8939_NEUROFEEDSTIM; 2017-A00809-44 (Other: ANSM); 17/051-1 (Other: CPP Ouest V (Rennes))
Record Dates: First submitted 2017-09-05; First posted 2017-09-12 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Depression
Keywords: Depression, neurofeedback, TMS
MeSH Terms: conditions — Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EEG-neurofeedback training in association with TMS. (Experimental): EEG-neurofeedback training in association with TMS.
  Interventions: Device: EEG-neurofeedback training in association with TMS.

INTERVENTIONS:
Device: EEG-neurofeedback training in association with TMS. — EEG-neurofeedback training in association with TMS.

SUMMARY:
Neurofeedback is an increasingly researched technique for the treatment of many psychological disorders, such as attention deficit / hyperactivity disorder (AD / HD), depression, or substance abuse. This technique would allow patients to regulate their cortical electroencephalographic activity while receiving a visual or auditory feedback on the cortical electroencephalographic activity. Changes in the electroencephalogram (EEG) would thus be correlated with changes in cortical activity and thus with symptoms.

On the electroencephalographic plane, the depression appears associated with relatively more alpha activity (in "resting state", 8-13 Hz) in left than in right frontal cortex. This difference in alpha activity between frontal regions is known as alpha asymmetry in depression. As a reminder, increased alpha activity indicates a decrease in cortical activation. This alpha asymmetry appears to be associated with a decrease in sensitivity to reward.

It is on these bases that the modification of the alpha asymmetry has become one of the most frequent objectives of the studies on the use of neurofeedback in depression.

Transcranial magnetic stimulation (TMS) also offers a non-invasive and painless method of effective cerebral stimulation in psychiatric disorders and especially depression. It received a favorable opinion from the Food & Drug Administration (FDA) in the United States for the treatment of this pathology. This treatment is still under evaluation in France. The results are promising but improvements must be done to increase its effectiveness.

TMS offers stimulation of brain tissue in a localized and non-invasive manner. The principle consists of a brief electric current passing through a coil which generates a transient magnetic field inducing an electric field through conductive fabrics. TMS modifies neuronal activity in target superficial brain structures, but also modulates neuronal circuit activity.

In recent years, the concept of "state dependency TMS" has been developed. It suggests that the activation state of neuronal circuits before and after stimulation alters the effect of stimulation. Thus, the efficacy of TMS could be amplified in depression by taking into account the cerebral activity during the stimulation sessions, in particular on the electroencephalographic plane.

However, TMS may also help patients increase their EEG response during Neurofeedback sessions.

The combination of stimulation techniques and brain-machine interfaces such as neurofeedback is still little studied at present.

A study on the combined use of TMS and Neurofeedback by EEG in depression would therefore be an innovative approach and in line with the latest data from the literature.

Design : Prospective, monocentric, non-randomized, non-comparative, unblinded study.

DETAILED DESCRIPTION:
Primary objective : To demonstrate a decrease in the intensity of depressive symptomatology following EEG-neurofeedback training in association with TMS and see if there is a correlation with a change in frontal asymmetry.

Secondary objective : To demonstrate a cognitive improvement in patients with respect to motivation and control of thoughts, as well as perceived health, self-esteem and anxiety following EEG-neurofeedback training in association with TMS and to see if there is a correlation between the change in scores on psychometric scales with a change in frontal asymmetry.

The expected outcomes of this study are:

* Better characterization of the pathophysiological processes involved in depressive disorder;
* An evaluation of the effectiveness of EEG-Neurofeedback training in recurrent depressive disorder in association with TMS, both emotionally and cognitively;
* The development of innovative technologies in the field of brain-machine interfaces and optimization of procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a major depressive episode (DSM IV-TR 296) with an indication of TMS (whether or not they have previously benefited from TMS);
* Aged 18 and over;
* With a score greater than or equal to 15 at the MADRS;
* Under stable and unchanged pharmacological treatment for at least one month;
* Having signed a free and informed consent to participate in the study.

Non inclusion Criteria:

* Other psychiatric disorder of axis 1 of DSM IV-TR (schizophrenia, substance abuse / dependence, ...);
* Neurological or dementia history according to DSM criteria;
* Pregnant or nursing women;
* Major persons subject to legal protection (safeguard of justice, curators, guardianship);
* Participation in another research involving the human interventionist or at risk and minimal constraints
* Confined hospitalized patients (SDT, SDRE).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2018-09-07 (Actual); Study Completion 2019-09-07 (Actual)

PRIMARY OUTCOMES:
MADRS score | Baseline and day 12
  Total score at the MADRS (Montgomery and Asberg Depression Scale) scale: difference between day 1 and day 12.

SECONDARY OUTCOMES:
MADRS score | Day 1, day 12 and month 1
  Difference at the MADRS score between day 1, day 12 and month 1
BDI score | Day 1, day 12 and month 1
  Difference at the BDI score between day 1, day 12 and month 1
HAM-A score | Day 1, day 12 and month 1
  Difference at the HAM-A score between day 1, day 12 and month 1
TCAQ score | Day 1, day 12 and month 1
  Difference at the TCAQ score between day 1, day 12 and month 1
BIS-BAS system score | Day 1, day 12 and month 1
  Difference at the BIS-BAS system score between day 1, day 12 and month 1
SES score | Day 1, day 12 and month 1
  Difference at the SES score between day 1, day 12 and month 1
MHLCS score | Day 1, day 12 and month 1
  Difference at the MHLCS score between day 1, day 12 and month 1
Neuropsychological test | Day 1, day 12 and month 1
  Difference at the neuropsychological performance between day 1, day 12 and month 1
Frontal asymmetry alpha measurement. | Day 1, day 12 and month 1
  Difference at the frontal asymmetry alpha between day 1, day 12 and month 1

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Drapier, MD, Principal Investigator — Centre Hospitalier Guillaume Regnier
Locations (1):
- Centre Hospitalier Guillaume Régnier, Rennes, Britanny, France

IPD SHARING:
Plan to Share IPD: No